CLINICAL TRIAL: NCT00283192
Title: A Randomized, Double-Blinded, Placebo Controlled, Trial of the Effect of Sertraline Vs. Placebo in Reducing the Incidence and Severity of Hot Flashes in Healthy Women
Brief Title: Flushes and Sertraline Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H5287-23467-03; FAST
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2006-08-04 (Estimated); Status verified 2005-08

CONDITIONS: Menopause-Hot Flashes
Keywords: Menopausal Symptoms; Hot flashes
MeSH Terms: conditions — Hot Flashes | interventions — Sertraline

INTERVENTIONS:
Drug: Sertraline

SUMMARY:
The primary outcome of FAST (a randomized double-blinded, placebo controlled, trial of the effect of sertraline vs. placebo in reducing the incidence and severity of hot flushes in healthy women) is to determine if 6 weeks of treatment with sertraline (50mg daily for 2 weeks, followed by 100mg per day for 4 weeks, if tolerated) results in a greater reduction in hot flush score (frequency * severity) compared to placebo among women with moderate to severe hot flashes. The secondary aim is to determine the effect of treatment with sertraline on quality of life, sleep, sexual function, and mood.

DETAILED DESCRIPTION:
The primary aim of FAST is to determine if 6 weeks of treatment with sertraline (50 mg daily for 2 weeks, followed by 100 mg per day for 4 weeks, if tolerated) results in greater reduction in hot flush score (frequency x severity), frequency and severity compared to placebo among women with moderate to severe hot flushes.

The Secondary Aims:To determine the effect of treatment with sertraline on quality of life, sleep, sexual function, mood, and cognitive function. To determine if a modified, short version of a sexual function instrument is valid.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 - 60 years old
* Report > 14 hot flushes per week
* Willing to be randomized to sertraline or placebo
* Sign informed consent

Exclusion Criteria:

* History of bilateral oophorectomy
* Breast or ovarian cancer
* Liver disease
* Kidney disease requiring dialysis
* History of major depression (reported history of depression requiring therapy, hospitalization for depression, taking antidepressant drugs, history of suicide attempt)
* History of bipolar affective disorder (reported history of bipolar disorder requiring therapy, medications, hospitalized for bipolar disorder)
* Seizure disorder
* History of hypersensitivity to sertraline or to SSRIs
* Pregnancy or breast feeding
* Any medical or psychiatric condition which, in the investigator's opinion, would preclude the participant from adhering to the protocol or completing the trial;
* No estrogens or progestins for 3 months prior to screening or during enrollment
* Selective estrogen receptor modulators (SERMS)
* The following medications: clonidine, gabapentin, tricyclic antidepressants, monoamine oxidase (MAO) inhibitors, selective serotonin reuptake inhibitors (SSRIs), megesterol , oral contraceptives, androgens; and medications that are listed on the Pfizer Pharmaceutical drug insert as "contraindicated"

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100
Dates: Start 2003-07; Study Completion 2006-01

PRIMARY OUTCOMES:
To determine if 6 weeks of treatment with sertraline (50 mg daily for 2 weeks, followed by 100 mg per day for 4 weeks, if tolerated) results in greater reduction in hot flush score (frequency x severity), frequency and severity compared to placebo

SECONDARY OUTCOMES:
To determine the effect of treatment with sertraline on quality of life, sleep, sexual function, and mood. To determine if a modified, short version of a sexual function instrument is valid.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah G Grady, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Women's Health Clinical Research Center, San Francisco, California, United States

REFERENCES:
- [Derived] Grady D, Cohen B, Tice J, Kristof M, Olyaie A, Sawaya GF. Ineffectiveness of sertraline for treatment of menopausal hot flushes: a randomized controlled trial. Obstet Gynecol. 2007 Apr;109(4):823-30. doi: 10.1097/01.AOG.0000258278.73505.fa. PMID 17400842